CLINICAL TRIAL: NCT02124083
Title: Phase 1/2 Study of Vorinostat Therapy in Niemann-Pick Disease, Type C1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Washington University School of Medicine (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140102; 14-CH-0102 (Other: The National Institutes of Health)
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01-13

CONDITIONS: Neimann-Pick Disease
Keywords: Niemann Pick Disease, Type C1; Phase I, Phase 2; Vorinostat
MeSH Terms: conditions — Niemann-Pick Disease, Type A; Niemann-Pick Disease, Type C | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vorinostat (Experimental): Trial participants were treated with Vorinostat (3 days on/4 days off regimen) to limit toxicity. Subjects were initially dosed with 200 mg (two 100 mg capsules) by mouth daily for three months, followed by dose escalation to 400 mg (four 100 mg capsules) by mouth daily for three months.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Histone deactylase inhibitor

SUMMARY:
Niemann-Pick disease type C (NPC) is a lethal, autosomal recessive, lysosomal storage disorder characterized by neurodegeneration in early childhood and death in adolescence. The causative genes NPC1 (about 95% of cases) and NPC2 (about 5% of cases) are involved in the intracellular trafficking of lipids and cholesterol. Mutations on either of these genes lead to progressive accumulation of unesterified cholesterol and other lipids in the central nervous system (CNS). Vorinostat is a histone deacetylase inhibitor that has been shown in vivo to increase mutant NPC1 protein levels and to reverse cellular accumulation of unesterified cholesterol. Vorinostat has been labeled by the FDA for treatment of cutaneous T-cell lymphoma. In this Phase I, non-randomized, open-label, single-center study, we plan to study whether Vorinostat can be repurposed to treat patients with NPC1. Our primary objective is to determine the safety and tolerability of Vorinostat in NPC1 disease. Our secondary objectives will be to determine biochemical efficacy of Vorinostat to increase expression of NPC1 protein and normalize lipid and protein biomarkers. This study will enroll up to 12 NPC1 patients and test the safety of two dose levels (200 and 400 mg). Drug will be administered on a 3 days on/4 days off schedule for 3 months at each dose level. Patients will be evaluated at the NIH Clinical Center at 0, 3 and 6 months. Safety will be assessed by adverse events (AEs), clinical laboratory tests and physical examinations. Biochemical efficacy will be assessed by measurement of serum and cerebral spinal fluid biomarkers. Clinical efficacy will be evaluated by audiologic testing, assessment ataxia, and swallowing studies.

DETAILED DESCRIPTION:
Niemann-Pick disease type C (NPC) is a lethal, autosomal recessive, lysosomal storage disorder characterized by neurodegeneration in early childhood and death in adolescence. The causative genes NPC1 (about 95% of cases) and NPC2 (about 5% of cases) are involved in the intracellular trafficking of lipids and cholesterol. Mutations on either of these genes lead to progressive accumulation of unesterified cholesterol and other lipids in the central nervous system (CNS). Vorinostat is a histone deacetylase inhibitor that has been shown in vivo to increase mutant NPC1 protein levels and to reverse cellular accumulation of unesterified cholesterol. Vorinostat has been labeled by the FDA for treatment of cutaneous T-cell lymphoma. In this Phase I, non-randomized, open-label, single-center study, we plan to study whether Vorinostat can be repurposed to treat patients with NPC1. Our primary objective is to determine the safety and tolerability of Vorinostat in NPC1 disease. Our secondary objectives will be to determine biochemical efficacy of Vorinostat to increase expression of NPC1 protein and normalize lipid and protein biomarkers. This study will enroll up to 12 NPC1 patients and test the safety of two dose levels (200 and 400 mg). Drug will be administered on a 3 days on/4 days off schedule for 3 months at each dose level. Patients will be evaluated at the NIH Clinical Center at 0, 3 and 6 months. Safety will be assessed by adverse events (AEs), clinical laboratory tests and physical examinations. Biochemical efficacy will be assessed by measurement of serum and cerebral spinal fluid biomarkers. Clinical efficacy will be evaluated by audiologic testing, assessment ataxia, and swallowing studies.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Aged greater than or equal to 18 and less than or equal to 60 years old at time of enrollment, either gender, and any ethnicity.
2. Diagnosis of NPC1 based upon one of the following:

   * Two NPC1 mutations;
   * Positive filipin staining and at least one NPC1 mutation;
   * Vertical supranuclear gaze palsy (VSNGP) in combination with either:
   * One NPC1 mutation, or
   * Positive filipin staining and no pathogenic NPC2 mutations.
3. Patients with at least one neurological manifestation of NPC1. For example, but not limited to, hearing loss, vertical supranuclear gaze palsy, ataxia, dementia, dystonia, seizures, dysarthria, or dysphagia.
4. A patient s cultured skin fibroblasts when treated with 10 M Vorinostat must exhibit a reduction in the filipin lysosomal storage organelle ratio equivalent to 75% of the response measured in NPC1 positive control fibroblasts.
5. Ability to travel to the NIH Clinical Center repeatedly for evaluation and follow-up.
6. If taking miglustat, the patient must have been taking a constant dose of the medication for no less than three months prior to baseline evaluation and must be willing to maintain that dose level for the duration of the trial.
7. Willing to discontinue all non-prescription supplements, with the exception of an age-appropriate multivitamin.
8. Women of reproductive age must be willing to use an effective method of contraception for the duration of the trial.
9. Willing to participate in all aspects of trial design including serial blood and CSF collections.

EXCLUSION CRITERIA:

1. Aged below 18 or above 60 years of age at enrollment in the trial.
2. Severe manifestations of NPC1 that would interfere with the patient s ability to comply with the requirements of this protocol.
3. Neurologically asymptomatic patients.
4. Patients who have received any form of cyclodextrin or an HDACi in an attempt to treat NPC1.
5. History of hypersensitivity reactions to Vorinostat or components of the formulation.
6. Pregnancy or breastfeeding at any time during the study.
7. Patients with suspected infection of the CNS or any systemic infection.
8. Neutropenia, defined as an absolute neutrophil count (ANC) of less than 1,500 per microliter.
9. Thrombocytopenia defined as a platelet count less than 75,000 per microliter, or a history of greater than or equal to grade 2 thrombocytopenia (50,000-75,000 platelets/microliter).
10. Prior use of anticoagulants or history/presence of a bleeding disorder.
11. Hepatic laboratory parameters (aspartate aminotransferase (AST), alanine aminotransferase, (ALT)) greater than four-times upper limit of normal.
12. Presence of anemia defined as two standard deviations below normal for age and gender.
13. Serum creatinine level greater than 1.5 times the upper limit of normal.
14. Hematuria (greater than15 RBC/mcL or positive hemoglobin). This exclusion criteria will not apply to a female currently menstruating who has no history of renal disease or other evidence of renal impairment (eg hypertension, serum creatinine above upper limit of normal, history of renal disease). Urinalyis will be repeated after menses has ended and drug discontinued if hematuria persists. Efforts will be made to avoid menses in scheduling the initial admission.
15. Proteinuria (1+ protein on urinalysis) Patient will not be excluded if urine protein/creatinine ratio is normal or if classified as benign by either patient's primary medical provider or upon obtaining a nephrology consult.
16. Serum potassium or Magnesium outside of the normal laboratory range prior to initiation of vorinostat therapy.
17. Diabetes or a fasting glucose greater than 106 mg/dl.
18. Active pulmonary disease, oxygen requirement or clinically significant history of decreased blood oxygen saturation, pulmonary therapy, or requiring active suction.
19. Patients with uncontrolled seizures per either of the criteria below.

    1. Unstable frequency, type or duration of seizures. Quantified by a seizure log over the two months prior to enrollment.
    2. Patients requiring antiepileptic medication changes (other than dose adjustments for weight) in the two months prior to enrollment, or requiring three or more antiepileptic medications to control seizures.
20. Use of another HDAC inhibitor or compounds with established HDAC inhibitory activity, including valproic acid, unless discontinued at least 2 months prior to enrollment.
21. History of a thromboembolic event (such as DVT or Pulmonary embolism).
22. Patients, who in the opinion of the investigators, are unable to comply with the protocol or have specific health concerns that would potentially increase the risk of participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04-25; Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Vanier MT. Niemann-Pick diseases. Handb Clin Neurol. 2013;113:1717-21. doi: 10.1016/B978-0-444-59565-2.00041-1. PMID 23622394
- [Background] Ory DS. Niemann-Pick type C: a disorder of cellular cholesterol trafficking. Biochim Biophys Acta. 2000 Dec 15;1529(1-3):331-9. doi: 10.1016/s1388-1981(00)00158-x. No abstract available. PMID 11111100
- [Background] Sevin M, Lesca G, Baumann N, Millat G, Lyon-Caen O, Vanier MT, Sedel F. The adult form of Niemann-Pick disease type C. Brain. 2007 Jan;130(Pt 1):120-33. doi: 10.1093/brain/awl260. Epub 2006 Sep 26. PMID 17003072
- [Derived] Garcia AA, Koperniku A, Ferreira JCB, Mochly-Rosen D. Treatment strategies for glucose-6-phosphate dehydrogenase deficiency: past and future perspectives. Trends Pharmacol Sci. 2021 Oct;42(10):829-844. doi: 10.1016/j.tips.2021.07.002. Epub 2021 Aug 10. PMID 34389161
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-CH-0102.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorinostat
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Secondary Outcome: Biochemical Efficacy as Measured by Serum Cathepsin D
Description: Serum concentration of Cathepsin D. Cathepsin D is an aspartyl protease involved in protein catabolism and tissue remodeling. Cathepsin D normal range = 220-515 ng/ml.
Time Frame: 6 months
Population: All participants completing both 200 and 400 mg phases
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vorinostat
Number analyzed (Participants) | 11
ng/mL | 625.3 (183.8)

2. Secondary Outcome: Biochemical Efficacy as Measured by Serum Cathepsin D
Description: as for outcome 1
Time Frame: Baseline
Population: All participants who started study
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vorinostat
Number analyzed (Participants) | 12
ng/mL | 648.2 (266)

3. Secondary Outcome: Biochemical Efficacy as Measured by Serum LGALS3
Description: Serum concentration of LGALS3 (galectin-3). Galectin-3 is a carbohydrate-binding lectin whose expression is associated with inflammatory cells including macrophages, neutrophils, and mast cells. LGALS3 normal range = 1.4-5.3 ng/ml.
Time Frame: 6 months
Population: All participants completing both 200 and 400 mg phases
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vorinostat
Number analyzed (Participants) | 11
ng/mL | 6.565 (4.775)

4. Secondary Outcome: Biochemical Efficacy as Measured by Serum LGALS3
Description: as for outcome 3
Time Frame: Baseline
Population: All participants who started study
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vorinostat
Number analyzed (Participants) | 12
ng/mL | 6.667 (2.303)

5. Primary Outcome: Number of Participants With Tolerabilty of 200 mg Vorinostat in Niemann-Pick Disease, Type C1
Description: The number of Niemann-Pick Disease, type C1 patients completing 3 month 200 mg phase
Time Frame: 3 months
Population: All participants who started study
Measure: Number; unit: Participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 12
Participants | 12

6. Primary Outcome: Number of Participants With Tolerabilty of 400 mg Vorinostat in Niemann-Pick Disease, Type C1
Description: The number of Niemann-Pick Disease, type C1 patients completing 3 month 400 mg phase
Time Frame: 3 months
Population: All participants completing 200 mg phase and starting 400 mg phase
Measure: Number; unit: Participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vorinostat
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat (N=12)
Vomiting (Gastrointestinal disorders) | 1
Epstein-Barr viraemia (Infections and infestations) | 1
Pyrexia (Infections and infestations) | 1
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 2
Liver function test increased (Investigations) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat (N=12)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastrostomy tube site complication (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Irritability (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Lip infection (Infections and infestations) | 1
Mouth ulceration (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Liver function test increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 4
Cataplexy (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Tracheostomy (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No